CLINICAL TRIAL: NCT05087342
Title: A Randomized Latino Semaglutide 2.4mg Study
Brief Title: Latino Semaglutide Study
Acronym: LSS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Loma Linda University (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Principal Investigator, Warren Peters, MD, MPH, Medical Director, Center for Health Promotion, Loma Linda University and Associate Professor, School of Medicine, Loma Linda University, Loma Linda University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 5210364
Record Dates: First submitted 2021-09-20; First posted 2021-10-21 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Obesity; Obesity; Drug; Overweight or Obesity; Weight Loss; Weight Loss Trajectory; Weight, Body
Keywords: obesity; obesity; drug; overweight; weight loss; weight
MeSH Terms: conditions — Obesity; Overweight; Weight Loss; Body-Weight Trajectory; Body Weight | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intervention Group (Active Comparator): Will receive active medication semaglutide subcutaneously, once weekly, self-injection.
  Month 1 - 0.24 mg SC once weekly x 4 weeks.(IE-1) Month 2- 0.5 mg SC once weekly x 4 weeks.(IE-2) Month 3 -1 mg SC once weekly x 4 weeks.(IE-3) Month 4 - 1.7 mg SC once weekly x 4 weeks.(IE-4) Month 5 - 2.4 mg SC once weekly x 4 weeks. (IE-5) Month 6 - 2.4 mg SC continue once weekly x 8 weeks.(IE-6) Month 7 - completion visit (IE-7)
  Interventions: Drug: Semaglutide 2.4mg
- Control Group (Placebo Comparator): Will receive placebo, subcutaneously, once weekly, self-injection throughout study duration.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Semaglutide 2.4mg — The intervention drug, semaglutide 2.4mg will be given to the Intervention Group per the schedule outlined in the armed description.
  Arms: Intervention Group
Drug: Placebo — A placebo will be given to the control group per the schedule outlined in the armed description.
  Arms: Control Group

SUMMARY:
The purpose of this study to understand better how this anti-obesity medication works to assist individuals to lose weight and maintain weight loss. This study may lead to the development of other related medications for assisting people with the disease of obesity.

ELIGIBILITY:
Inclusion Criteria:

* Self-identify as being of Hispanic/Latino ethnicity
* BMI >30
* Age 18-75 years old
* Able to provide informed consent before any trial related activities

Exclusion Criteria:

* Current cancer treatment
* Diabetes, Type 1 or Type 2
* Eating disorders
* Medication use targeting the GPL-1 system
* In the last 30 days, attempted to lose weight by lifestyle modification alone or with the use of anti-obesity medications resulting in more than 5 pounds of weight loss.
* History of bariatric surgery
* Use of obesogenic medications (including but not limited to steroids, haloperidol, clozapine, risperidone, olanzapine, amitriptyline, imipramine, paroxetine, and lithium) which cannot be substituted or stopped.
* Pregnant or planning to become pregnant in the next 8 months
* Genetic disorders and/or physical or mental handicaps that would limit participation in the study and/or the intensive lifestyle intervention.
* Any contraindication to semaglutide 2.4 mg including personal or family history of medullary thyroid carcinoma or Multiple Endocrine Neoplasia Syndrome Type 2, hypersensitivity to semaglutide 2.4 mg or any product components.
* Any known or suspected allergy to semaglutide 2.4 mg or related products
* Previous participation in this trial, either initial screening or group randomization

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2022-12-13 (Actual); Primary Completion 2024-05-29 (Actual); Study Completion 2024-05-29 (Actual)

PRIMARY OUTCOMES:
Assessment of weight loss. | Change between baseline and final study visit, seven months post baseline.
  Assessment will be based on pounds lost between baseline and final study visit.

SECONDARY OUTCOMES:
Food Addiction Assessment | Change between baseline and month four of treatment.
  Yale Food Addiction Scale Survey administered to subjects at baseline and month four of treatment. Assessment results based on multiple survey questions regarding intake of specific food types (sugar, starch, sweet, salty, savory).

CONTACTS AND LOCATIONS:
Overall Officials: Warren Peters, MD, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda University Health, Loma Linda, California, United States